CLINICAL TRIAL: NCT04147091
Title: Influence of Nano-hydroxyapatite and Ozone on Approximal Initial Caries
Brief Title: Nano-hydroxyapatite and Ozone - Effect on Approximal Initial Caries
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Pomeranian Medical University Szczecin (Other)
Responsible Party: Principal Investigator, Katarzyna Grocholewicz, Prof. DDS, PhD, Pomeranian Medical University Szczecin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KB-0012/102/11
Record Dates: First submitted 2019-10-21; First posted 2019-10-31 (Actual); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: Caries,Dental
MeSH Terms: conditions — Dental Caries | interventions — Wound Healing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- domestic nanohydroxyapatite gel ApaCare & Repair (Experimental): 6-months treatment, caries lesions were assessed on bitewing radiographs at baseline, after 1 year and after 2 years
  Interventions: Other: ApaCare & Repair
- in-office ozone therapy OzonyTron (Experimental): 6-months treatment, caries lesions were assessed on bitewing radiographs at baseline, after 1 year and after 2 years
  Interventions: Other: ApaCare & Repair
- both remineralizing gel and ozone therapy (Experimental): 6-months treatment, caries lesions were assessed on bitewing radiographs at baseline, after 1 year and after 2 years
  Interventions: Other: ApaCare & Repair

INTERVENTIONS:
Other: ApaCare & Repair — Initial cariuos lesions were treated.
  Other Names: OzonyTron

SUMMARY:
Objectives: to assess the efficiency of three methods of enamel remineralization on initial approximal caries: 1. a nano-hydroxyapatite gel, 2. gaseous ozone therapy 3. combination of a nano-hydroxyapatite gel and ozone.

Materials and Methods: Patients (n=92, age 20-30y) with initial approximal enamel lesions on premolar and molar teeth (n=546) randomly allocated to three groups subjected to a 6-months treatment: Group I: domestic nano-hydroxyapatite remineralizing gel, group II: in-office ozone therapy, group III: both remineralizing gel and ozone therapy. Caries lesions assessed on bitewing radiographs at baseline, after 1 year and after 2 years.

ELIGIBILITY:
Inclusion Criteria:

-initial approximal enamel lesions on premolar and molar teeth

Exclusion Criteria:

* distal surface of the last tooth in arch, overlapping teeth
* fillings on approximal surfaces of teeth of interest
* ongoing orthodontic therapy with braces or other appliances

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2012-02 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Remineralizing effect | baseline
  Caries lesions were assessed on bitewing radiographs

SECONDARY OUTCOMES:
Remineralizing effect - follow-up | after 1 year and after 2 years
  Caries lesions were assessed on bitewing radiographs